CLINICAL TRIAL: NCT04346498
Title: The Effect of Chest-to-Back Skin-to-Skin Contact on Regulation of Physiological Parameters for Low Birth Weight and/or Premature Infants: a Crossover Randomized Controlled Clinical Trial
Brief Title: Can Kangarooing Small Babies on the Back of a Mother Keep Them Warm and Stable
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SISAY GERE (Other)
Collaborators: Arsi University (Other); Adds Continental Institute of Public Health (Unknown)
Responsible Party: Sponsor-Investigator, SISAY GERE, MSc, PhD candidate, and lecturer at Arsi University College of Health Sciences, Ethiopia, Addis Continental Institute of Public Health
Organization: Addis Continental Institute of Public Health (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A/CHS/RC/15/16
Record Dates: First submitted 2020-04-11; First posted 2020-04-15 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Body Temperature; Oxygen Saturation; Heart Rate; Respiratory Rate; Sleep Pattern

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Mothers were masked only for the presence or absence of a sequence in the trial. Hospital staffs, students, and investigators of the study were all blinded to allocation of the intervention. Until the study was finalized, access to the database was restricted to the data manager only
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CB-SSC (Experimental): The participant received CB-SSC for 2 hours per day for three consecutive days
  Interventions: Other: Chest-to-back
- CC-SSC (Placebo Comparator): Following a 30 minute washout time, the same participant would continue to receive chest-to-chest (CC) SSC for 2 hours. This was also conducted for three consecutive days
  Interventions: Other: Chest-to-back

INTERVENTIONS:
Other: Chest-to-back
  Other Names: The standard/or Chest-to-chest

SUMMARY:
The purpose of this study was to assess the effectiveness of Kangarooing small babies on the back of a mother

DETAILED DESCRIPTION:
After the study was explained (risks and benefits) and written informed consent was received from participants, an individually controlled randomized crossover clinical trial was conducted to examine the effectiveness of Chest-to-Back (CB) skin-to-skin contact (SSC) compared with the standard. The trial was done in accordance with the protocol, good clinical practice, and the national regulatory and ethics guideline of Ethiopia (which is in line with the Helsinki declaration).

ELIGIBILITY:
Inclusion Criteria:

* Neonates with LBW (<2500 grams)
* Born prematurely (< 37 complete weeks of gestation)

Exclusion Criteria:

* less than 35 weeks of gestation on the day of enrollment to trial
* Malformations or birth disabilities
* Dependent on oxygen or IV fluid
* Any disorder that was deemed necessary for exclusion by the investigator.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-10-14 (Actual)

PRIMARY OUTCOMES:
Change in skin temperature from baseline | : From the start of SSC (0 hour) to end of SSC (2 hours) per day, assessed for three consecutive days
  Skin temperature values were recorded every 10 minutes. Including the baseline, the 2 hours intervention would provide 13 measurements. A participant who successfully completed the intervention would have78 measurements; 39 for the treatment arm and 39 for the control arm.

OTHER OUTCOMES:
Change from baseline in peripheral arterial oxygen saturation on SCRIP Score | From the start of SSC (0 hour) to end of SSC (2 hours) per day, assessed for three consecutive days
  Stability of the cardio-respiratory system in premature infants (SCRIP) score is a reliable instrument for determining the stability of oxygen saturation (i.e., peripheral arterial oxygen saturation) in premature infants. Possible scores range from 2 (perfect stability= > 90 %) to 0 (sever instability = any falls below 80%)
Change from baseline in heart rate on SCRIP Score | From the start of SSC (0 hour) to end of SSC (2 hours) per day, assessed for three consecutive days
  Possible scores range from 2 (perfect stability= regular) to 0 (sever instability = < 80/min or>200).
Change from baseline in respiratory rate on SCRIP Score | From the start of SSC (0 hour) to end of SSC (2 hours) per day, assessed for three consecutive days
  Possible scores range from 2 (perfect stability= regular) to 0 (sever instability = Apnea> 10, Tachypnea> 80/min, fussing/agitation
Length of sleep in minute | From the start of SSC (0 hour) to end of SSC (2 hours) per day, assessed for three consecutive days.
  length of sleep was defined by the duration between the time of closed eyes, no crying and no movement to the time that at least one of these 3 indicators is absent

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Yemane Berhane, Study Director — Director; Prof. Alemayehu Worku, Study Chair — Deputy
Locations (1):
- Adds Continental Institute of Public Health, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
Upon a reasonable request, the investigators can offer access to the datasets used and/or analyzed. This can be available from the PI (principal investigator)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Possibly after six months the data will be available.
Access Criteria: Upon reasonable request!